SAP, 43CH1626, Restylane Volyme Midface

NCT03289052

MA-35135

2022-12-09 10:56

Print date:

Effective date: 2017-11-03 11:43



**Clinical Trial Number: 43CH1626** 

A randomized, multi-center, evaluator-blinded, no-treatment controlled study to evaluate the effectiveness and safety of Restylane Volyme for correction of Midface Volume Deficit and/or Midface Contour Deficiency 👶 GALDERMA

SAP, 43CH1626, Restylane Volyme Midface

Doc id

Print date:

MA-35135

# **Table of Contents**

| 1 | Stud | y Information | 3 |
|---|---|---|---|
| | 1.1.1 | Study design | ŝ |
| | 1.1.2 | Number of subjects and randomization | ŝ |
| | 1.2 | Study Objectives | 3 |
| | 1.3 I | Effectiveness Assessments | 4 |
| | 1.3.1 | Medicis Midface Volume Scale (MMVS) | 4 |
| | CCI | | 4 |
| | | ······································ | 4 |
| | | | 5 |
| | 1.4 I | Effectiveness Endpoints | 5 |
| | 1.4.1 | Primary effectiveness endpoint | 5 |
| | CCI | | 5 |
| | 1.5 | Safety Assessments | <i>6</i> |
| | 1.6 | Safety Endpoints | 7 |
| 2 | Stati | stical Methods | 7 |
| | 2.1 | General Methods | 7 |
| | 2.2 A | Analysis Populations | 8 |
| | 2.3 | Study Subjects | 8 |
| | 2.3.1 | Subject disposition | 8 |
| | 2.3.2 | Protocol deviations | 9 |
| | 2.3.3 | Demographics and Baseline characteristics | 9 |
| | 2.3.4 | Medical history, and concomitant medication and procedures | 10 |
| | 2.3.5 | Extent of exposure | 10 |
| | 2.3.6 | Post-treatment examinations | 11 |
| | 2.4 I | Effectiveness Analysis | 11 |
| | 2.4.1 | Data sets analyzed | 11 |
| | 2.4.2 | Handling of missing data | 11 |
| | 2.4.3 | | |
| | CCI | | 12 |
| | | Safety Analysis | |
| | CCI | | 13 |
| | 2.5.2 | Adverse Events | 13 |

| • GALDERMA | SAP, 43CH1626, Restylane Volyme Midface |
|------------|-----------------------------------------|

Doc id

# MA-35135

| | 2.6 | Interim Analysis | 14 |
|---|-----|----------------------------------------------------|-----------|
| | 2.7 | Determination of Sample Size | 14 |
| | 2.8 | Changes in the Analysis Planned in the Protocol | 14 |
| 3 | I | Reference List | 15 |
| 4 | A | Appendix A1: Study Subjects | 16 |
| | 4.1 | Analysis Populations | 16 |
| | 4.2 | Protocol Deviations | 16 |
| | 4.3 | Subject disposition | 18 |
| 5 | A | Appendix A2: Demographics | 24 |
| | 5.1 | Demographics and baseline characteristics | 24 |
| | 5.2 | Medical history | 26 |
| 6 | A | Appendix A3: Concomitant medication and procedures | 29 |
| | 6.1 | Concomitant medication | 29 |
| | 6.2 | Concomitant procedures | 31 |
| 7 | A | Appendix A4: Treatment procedure | 32 |
| 8 | A | Appendix A5: Post-treatment examinations | 35 |
| 9 | A | Appendix A6: Effectiveness Evaluation for Group B | 36 |
| | 9.1 | Primary analysis | 36 |
| | 9 | 9.1.1 MMVS responder rate at Month 6 | 36 |
| | CCI | | 38 |
| | | | 39 |
| | | | 39 |
| | | | 45 |
| | | | 46 |
| | | | 48 |
| | | | 50 |
| 1 | | Appendix A7: Safety evaluation | <b>56</b> |
| | CCI | | |
| | 10. | 2 Adverse Events | 59 |
| | 1 | 10.2.1 Summary of Adverse Events (AEs) | 59 |
| | 1 | 10.2.2 Related AEs | 60 |
| | 1 | 10.2.3 Unrelated AFs | 63 |

SAP, 43CH1626, Restylane Volyme Midface

Doc id

Print date:

MA-35135

2022-12-09 10:56

Effective date: 2017-11-03 11:43

#### 1 **Study Information**

#### 1.1.1 Study design

This is a randomized, evaluator-blinded, no-treatment controlled study to evaluate the effectiveness and safety of Restylane Volyme for correction of Midface Volume Deficit and/or Midface Contour Deficiency in subjects of Chinese origin, men or women aged 18 years or older.

The study will be conducted at approximately 5 sites located in China, and subjects with a Medicis Midface Volume Scale (MMVS) score of 2, 3 or 4 on each side of the face, as assessed by the Blinded Evaluator, will be enrolled. The subjects will be followed for approximately 14 months.

Only the Evaluator will be blinded, both Treating Investigator and subjects will be aware of the treatment. To avoid inter-observer variability, every effort should be made to ensure that preferably the same individual who made the initial baseline determinations completes all corresponding follow-up evaluations.

For more details regarding the study, and references, please see the Clinical Study Protocol (CSP), MA-33281.

#### 1.1.2 Number of subjects and randomization

A total of approximately 168 subjects will be enrolled.

Up to 20 subjects (2 first treated subjects per Treating Investigator, with maximum 2 treating investigators per site) will be enrolled as group A and all subjects in this group will receive treatment with Restylane Volyme. In group B, approximately 148 subjects will be randomized ratio to treatment with Restylane Volyme or no treatment. The randomization will be stratified by site.

#### 1.2 **Study Objectives**

The study objectives are:

- To evaluate the effectiveness of Restylane Volyme in the treatment of Midface Volume Deficit and/or Midface Contour Deficiency.
- To evaluate the safety of Restylane Volyme in the treatment of Midface Volume Deficit and/or Midface Contour Deficiency.



### 1.3 Effectiveness Assessments

### 1.3.1 Medicis Midface Volume Scale (MMVS)

MMVS is a four-point photographic scale that assesses the fullness of the midface from 'Fairly full' (1) to 'Substantial loss of fullness' (4) as described below, see Table 1-1.



The Blinded Evaluator will rate the subject's right and left midface for severity of volume deficiency using the MMVS at screening, baseline, , 6, CCI months after last treatment in Group A and Treatment Group; and at screening, baseline, and 6 months after randomization, as well as and 6 months after last treatment in Control Group.





## 1.4 Effectiveness Endpoints

### 1.4.1 Primary effectiveness endpoint

The primary effectiveness endpoint is the percentage of responders, defined by at least 1 point improvement from baseline on the MMVS on both sides of the face concurrently, as measured by the Blinded Evaluator at 6 months after last treatment in Treatment Group and 6 months after randomization in Control Group.

| CCI |
|-----|

Print date: 2022-12-09 10:56 Doc id SAP, 43CH1626, Restylane Volyme Midface GALDERMA MA-35135

## 1.5 Safety Assessments



A two-point scale ('Yes' or 'No') will be used to assess causality of AEs, serious as well as non-serious. The Investigator shall be asked to indicate a response to each of the following questions in the electronic case report form (eCRF):

- "Do you consider that there is a reasonable possibility that the event may have been caused by the study product?" and
- "Do you consider that there is a reasonable possibility that the event may have been caused by the study product injection procedure?"

If any of these questions are answered with a 'Yes', the AE will be considered related.



Each AE will also be assessed for causal relationship and seriousness by the Sponsor, in order to fulfill regulatory requirements. In case of a disagreement, the AE will be considered 'Related'.

Any device deficiencies discovered in relation to treatment at baseline and 4-week follow-up visits for the Treatment Group and treatment at 6 months after randomization and 4-week follow-up after 6-moth treatment for the Control Group will be recorded.

### 1.6 Safety Endpoints

Safety endpoints include:



(ii) Incidence, intensity, duration, and onset of adverse events (AEs) collected throughout the study.

### **2** Statistical Methods

#### 2.1 General Methods



Print date:

2022-12-09 10:56

### 2.2 Analysis Populations

The following populations for Group B will be defined:

| • | Safety | Includes all subjects in Group B who were treated with |
|---|--------|----------------------------------------------------------|
| | | Restylane Volyme or randomized to no-treatment group. |
| | | Subjects are analyzed based on the as treated principle. |

• Full Analysis Set (FAS) Includes all subjects in Group B who were treated with Restylane Volyme or randomized to no-treatment group. Subjects are analyzed according to the randomization assignment.

• Per Protocol (PP) Includes all subjects in FAS that comply to the protocol procedures with no deviations that can affect the evaluation of the primary variable.

The FAS population is the primary population for all effectiveness analyses. All safety analyses will be based on the Safety population.

Group A will be followed for safety evaluation throughout the whole study.

### 2.3 Study Subjects

#### 2.3.1 Subject disposition

The number and percentage of subjects in each study population (FAS, PP, and Safety) will be summarized by site (including subject number) and in total (Table 4-1). Study population variables will also be presented in a data listing.

The disposition of subjects, including reason for withdrawals, will be presented by site and in total (Table 4-4). Number of completed, missed, and withdrawn subjects, as well as subjects continuing in the study will be accounted for by visit and treatment group (Table 4-5 and Table 4-6). Subject accountability will also be presented in a flowchart (Figure 4-1 and Figure 4-2).

All withdrawn subjects will be listed individually, including site number, subject number, treatment group, date of treatment and withdrawal, reason for withdrawal and last visit performed (Table 4-7 and Table 4-8).

Reasons for screening failures will be summarized (Table 4-9).



#### 2.3.2 Protocol deviations

Subjects with CSP deviations will be presented by observed protocol deviation, number of subjects and number of deviations (Table 4-3). Depending on the seriousness of the deviation, the subject might be excluded from the PP population (Table 4-2), which shall be documented prior to database lock (DBL).

Definition of protocol deviations that will exclude subjects from the PP are defined (but not limited to) in Table 2-1 below.

Table 2-1: Protocol deviations

| | | Deviation |
|---|---|---|
| GENERAL | | |
| | | Visit out-of-window |
| | * | Follow-up at 6 months after last treatment performed earlier than 1 week before the scheduled visit or later than 2 weeks after the scheduled visit in Treatment Group. |
| | * | Follow-up at 6 months after randomization performed earlier than 1 week before the scheduled visit or later than 2 weeks after the scheduled visit in Control Group. |
| EFFECTIVENESS | | |
| | | MMVS assessed by Blinded Evaluator |
| | * | Not done for both sides of the face at 6 months after last treatment in Treatment Group, or at 6 months after randomization in Control Group. |
| | * | Pre-treatment MMVS not available for both sides of the face. |
| | * | More than 1 grade difference in baseline MMVS score between the two sides of the face. |
| OTHER | | |
| | | Inclusion/exclusion criteria |
| | * | Any inclusion criteria affecting primary effectiveness evaluation not met. |
| | * | Any exclusion criteria affecting primary effectiveness evaluation met. |

#### 2.3.3 Demographics and Baseline characteristics

Demographic endpoints and subject baseline characteristics will be presented by treatment group (Table 5-1) using descriptive statistics. Gender, ethnic origin, and baseline MMVS score (assessed by Blinded Evaluator and ) will be summarized as categorical end points using number and percentage of subjects. Age and baseline BMI will be summarized by number of subjects, mean, standard deviation, minimum, median, and maximum values.

### 2.3.4 Medical history, and concomitant medication and procedures

All summaries will be based on the Safety population. Concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary. Medical history will be coded according to medical dictionary for regulatory activities (MedDRA).

#### Medical history/concurrent disease

The number and percentage of subjects reporting medical history/concurrent diseases and the number of conditions will be summarized by System Organ Class (SOC) and in total, for all medical history during the whole study and ongoing at study start (Table 5-2 and Table 5-3).

Prior use of facial fillers or implants will be summarized by type of fillers/implants using number and percentage of subjects and number of events (Table 5-4). Prior use of other facial dermatological procedures will be summarized by type of procedure using number and percentage of subjects and number of events (Table 5-5).

#### **Concomitant medication and procedures**

The number and percentage of subjects reporting concomitant medication ongoing at study start, initiated during study and in total (Table 6-1) will be summarized. In addition, the number and percentage of subjects reporting concomitant medication, and the number of medications will be summarized by reason and in total (Table 6-2). Also, the number and percentage of subjects, and the number of medications, will be summarized by ATC code and in total, along with an ATC text description (Table 6-3).

Concomitant medication taken due to an AE will be summarized by ATC code (along with an ATC text description) and in total using number and percentage of subjects and number of medications, and by MedDRA coded AE and whether the AE is related or not (Table 6-4 and Table 6-5).

Concomitant procedures will be presented by reason and in total (Table 6-6), as well as by type of procedure (Table 6-7), using number and percentage of subjects and number of procedures.

#### 2.3.5 Extent of exposure

Volume injected (mL), for each treatment visit and in total will be presented by treatment group (Table 7-1) using number of subjects, mean, standard deviation, minimum, median, and maximum values. Depth of injection and injection method for each treatment visit will be summarized by treatment group using number and percentage of subjects (Table 7-1).

Local anaesthesia used and post-treatment care for each treatment visit will be summarized by treatment group using number and percentage of subjects (Table 7-2).

Print date:

2022-12-09 10:56

#### 2.3.6 Post-treatment examinations

Change from baseline in post-treatment BMI will be presented for subjects with a change in  $BMI \ge 2$  units, if applicable (Table 8-1).

### 2.4 Effectiveness Analysis

### 2.4.1 Data sets analyzed

All effectiveness variables will be analyzed using the FAS population. The primary analysis will be repeated using the PP population. If it is deemed necessary, other analyses will be repeated using the PP population.

### 2.4.2 Handling of missing data

Number of missing values will be summarized and reported as appropriate.

Different assumptions regarding the missing data will be used. For the primary effectiveness analysis, missing values in the FAS will be assumed to be missing due to lack of effect. Therefore missing data up to the Month 6 visit will be imputed using the baseline observation carried forward (BOCF) method. As an alternative approach, missing data will be assumed to be unrelated to treatment effect. To impute data under this assumption, missing data up to the Month 6 visit will be imputed using the hot deck method (Table 9-2). Both of these alternatives will estimate the effectiveness of the treatment policy (irrespective of use of disallowed treatments, procedures, or medications) rather than the true, clinical treatment effect.

To obtain an estimate of the true, clinical treatment effect, the primary effectiveness analysis will be performed using the PP population.

All other endpoints will be analyzed on available data, i.e. no imputations will be done.



Doc id SAP, 43CH1626, Restylane Volyme Midface ♣ GALDERMA MA-35135

#### 2.4.3 Primary analysis

The percentage of responders (a responder will be defined as a subject with at least 1 point improvement from baseline MMVS on both sides of the face concurrently) will be calculated for each group at Month 6 (after last treatment for Treatment group, and after randomization











#### 2.5 Safety Analysis

All safety variables will be summarized descriptively based on the Safety population.



#### 2.5.2 Adverse Events

All AEs will be coded according to MedDRA and summarized by System Organ Class (SOC) and Preferred Term (PT). All AE summaries defined below will be presented by treatment, i.e. no treatment at baseline vs. all treated subjects (at baseline and Month 6).

An overall summary of number and percentage of subjects with any AEs, including related/unrelated and serious AEs, and the number of events will be compiled (Table 10-5).

For related AEs, maximum intensity of the AE will be summarized (Table 10-6). The duration (Table 10-7) and time to onset (Table 10-8) of event will be summarized by SOC and PT using number of events, mean, standard deviation, minimum, median, and maximum statistics. Action taken due to a related AE will be summarized by SOC, and PT (Table 10-9) using number of events.

Number and percentage of subjects with unrelated AEs and number of events will be presented by SOC, PT and maximum intensity (Table 10-10).

Time to onset of an AE will be derived as the start date minus the date of the most recent treatment. If the start date is missing, it will be assumed that the AE started on the date of the most recent treatment.

Duration of an AE will be derived as the stop date minus the start date +1. If the start date is missing, it will be assumed that the AE started on the date of the most recent treatment. Missing stop date will not be imputed and therefore no duration will be calculated in these cases. Instead, the number of AEs that were ongoing at the end of the study will be given.



### 2.6 Interim Analysis

No interim analysis is planned.

## 2.7 Determination of Sample Size

There are no available clinical data for Restylane Volyme studied under conditions similar to the current study. However, based on what is seen in clinical studies of injectable fillers in the facial areas, it is reasonable to assume a response rate of at least 70% in the Restylane Volyme treatment group at Month 6. For the no treatment control group, response rates as high as 35% have been observed in Glogau et al<sup>1</sup>. Based on this, it was assumed that the response rate will be maximum 35% in the no-treatment control group at Month 6.



## 2.8 Changes in the Analysis Planned in the Protocol

## **3** Reference List

Glogau RG et al. A randomized, evaluator-blinded, controlled study of the efficacy and safety of small gel particle hyaluronic acid for lip augmentation. Dermatol Surg. 2012 Jul; 38(7 Pt 2):1180-92.

| | SAP, 43CH1626, Restylane Volyme Midface | Doc id |
|-------------------|------------------------------------------|----------|
| <b>♣</b> GALDERMA | erry to errozo, root, and voying trained | MA-35135 |

# 4 Appendix A1: Study Subjects

## 4.1 Analysis Populations

**Table 4-1: Analysis populations** 

| Cito | Crown | Subject | Sa | fety | FA | S | Р | ·P |
|-----------|-------|---------|----|------|----|---|---|----|
| Site | Group | number | n | % | n | % | n | % |
| Site 1 | Α | 1xx-1xx | | | | | | |
| Sile i | В | 1xx-1xx | | | | | | |
| Site 2 | Α | 2xx-2xx | | | | | | |
| Sile 2 | В | 2xx-2xx | | | | | | |
| Site 3 | Α | 3xx-3xx | | | | | | |
| Sile 3 | В | 3xx-3xx | | | | | | |
| Site 4 | Α | 4xx-4xx | | | | | | |
| Sile 4 | В | 4xx-4xx | | | | | | |
| Site 5 | Α | 5xx-5xx | | | | | | |
| Sile 3 | В | 5xx-5xx | | | | | | |
| Total (N) | | | | | | | | |

<sup>% =</sup> n/N\*100

## **4.2** Protocol Deviations

Table 4-2: Protocol deviations excluding subjects from PP population, Group B

| Protocol deviation | Number of subjects <sup>1)</sup> | Subject numbers |
|--------------------|----------------------------------|-----------------|
| Total | | |

<sup>1)</sup> The same subject may have been excluded from PP for more than one reason.

Table 4-3: Protocol deviations not excluding subjects from PP population, Group A and B

| Drotocol | Gro | ıp A | Gro | ир В | Total |
|---|---|---|---|---|---|
| Protocol deviation | Number of subjects <sup>1)</sup> | Subject<br>numbers | Number of subjects <sup>1)</sup> | Subject<br>numbers | Total Number of deviations |
| Total | | | | | |

<sup>1)</sup> A single subject may have reported several protocol deviations.

Print date:

2022-12-09 10:56

## 4.3 Subject disposition

Table 4-4: Disposition of all subjects

| Site | Group | | eened<br>ojects | Enro<br>subje | | Subject Subjects Subjects Subjects | | | Withdrawn subjects | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | numbers | n | % | n | % | n | % |
| Site 1 | Α | | | | | 1xx-1xx | | | | | | |
| Sile i | В | | | | | 1xx-1xx | | | | | | |
| Site 2 | Α | | | | | 2xx-2xx | | | | | | |
| Site 2 | В | | | | | 2xx-2xx | | | | | | |
| Cito 3 | Α | | | | | 3xx-3xx | | | | | | |
| Site 3 | В | | | | | 3xx-3xx | | | | | | |
| C:4- 4 | Α | | | | | 4xx-4xx | | | | | | |
| Site 4 | В | | | | | 4xx-4xx | | | | | | |
| Cito E | Α | | | | | 5xx-5xx | | | | | | |
| Site 5 | В | | | | | 5xx-5xx | | | | | | |
| Total (N) | | | | | | | | | | | | |

<sup>% =</sup> n/N\*100

Table 4-5: Subject accountability by visit: subjects randomized to treatment with Restylane Volyme, Group B

| Vioit | Number of subjects | | | |
|---|---|---|---|---|
| Visit | Completed | Missed | Withdrawals | Continuing in study |
| Baseline/initial treatment | | | | |
| 4W follow-up/optional touch-up | | | | |
| 4W follow-up after last treatment | | | | |
| 3M after last treatment | | | | |
| 6M after last treatment | | | | |
| 9M after last treatment | | | | |
| 12M after last treatment | | | | |

🞝 GALDERMA

SAP, 43CH1626, Restylane Volyme Midface

Doc id

Print date:

MA-35135

Table 4-6: Subject accountability by visit: subjects randomized to no-treatment control, group B

| Visit | | | Number of subject | ets |
|---|---|---|---|---|
| Visit | Completed | Missed | Withdrawals | Continuing in study |
| Baseline | | | | |
| 4W follow-up | | | | |
| 3M follow-up | | | | |
| 6M follow-up/treatment | | | | |
| 4W follow-up/optional touch-up | | | | |
| 4W follow-up after last treatment | | | | |
| 3M after last treatment | | | | |
| 6M after last treatment | | | | |

Doc id SAP, 43CH1626, Restylane Volyme Midface ♣ GALDERMA **MA-35135** 

Print date:

Figure 4-1: Subject accountability by visit in Group A



Doc id SAP, 43CH1626, Restylane Volyme Midface ♣ GALDERMA **MA-35135** 

Print date:

Figure 4-2: Subject accountability by visit in Group B



Print date: 2022-12-09 10:56

GALDERMA SAP, 43CH1626, Restylane Volyme Midface Doc id MA-35135

Table 4-7: Withdrawn subjects, Group A

| | Subject | Date o | f treatment | Last visit | Date of | |
|---|---|---|---|---|---|---|
| Site | number | Initial treatment | Optional touch-up treatment | performed | Date of<br>withdrawal | Reason for withdrawal |

Table 4-8: Withdrawn subjects, Group B

| | | Subject | Date | of treatment | Last visit | Date of | |
|---|---|---|---|---|---|---|---|
| Treatment group | Site | number | Initial<br>treatment | Optional touch-up treatment | performed | withdrawal | Reason for withdrawal |
| Restylane Volyme | | | | | | | |
| Control | | | | | | | |

Effective date: 2017-11-03 11:43 Version: 1.0

Table 4-9: Screening failures

| | Gro | up A | Gro | ир В | Total |
|---|---|---|---|---|---|
| Reason for screening failure | | Screening<br>number | Number of subjects | Number of subjects | |

Print date:

2022-12-09 10:56

## 5 Appendix A2: Demographics

## 5.1 Demographics and baseline characteristics

Table 5-1: Summary of demographics and baseline characteristics, Safety population

| | | | | Group B | |
|---|---|---|---|---|---|
| Characteristics | Parameter | Group A<br>N = xx | Restylane<br>Volyme<br>N = xxx | Control<br>N = xx | Total<br>N = xxx |
| Age (years) | N | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Minimum | | | | |
| | Maximum | | | | |
| Gender | | | | | |
| Female | n (%) | | | | |
| Male | n (%) | | | | |
| Ethnic origin | | | | | |
| Han Chinese | n (%) | | | | |
| Other <sup>1)</sup> | n (%) | | | | |
| Baseline BMI | N | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Minimum | | | | |
| | Maximum | | | | |
| Baseline MMVS score, Blinded Evaluator | | | | | |
| right side | | | | | |
| Score 2 | n (%) | | | | |
| Score 3 | n (%) | | | | |
| Score 4 | n (%) | | | | |
| | ) Specification of | Other: | 1 | 1 | 1 |

<sup>% =</sup> n/N\*100

<sup>1)</sup> Specification of Other: ..., ...,

Effective date: 2017-11-03 11:43

SAP, 43CH1626, Restylane Volyme Midface

Doc id

Print date:

MA-35135

2022-12-09 10:56

| | | | | Group B | |
|---|---|---|---|---|---|
| Characteristics | Parameter | Group A<br>N = xx | Restylane<br>Volyme<br>N = xxx | Control<br>N = xx | Total<br>N = xxx |
| left side | | | | | |
| Score 2 | n (%) | | | | |
| Score 3 | n (%) | | | | |
| Score 4 | n (%) | | | | |



 $% = \frac{1}{N} =$ 

Effective

SAP, 43CH1626, Restylane Volyme Midface

Doc id

Print date:

MA-35135

2022-12-09 10:56

## 5.2 Medical history

Table 5-2: Subjects reporting medical history/concurrent diseases and number of conditions by MedDRA System Organ Class (SOC) in Group A, Safety population

| Drimon, COC | | Tot | al | Ongoing at study start | | |
|---|---|---|---|---|---|---|
| Primary SOC | Subje | cts | Conditions | Subje | cts | Conditions |
| | n | % | n | n | % | n |
| Total (N)1) | | | | | | |

<sup>% =</sup> n/N\*100

Effective date: 2017-11-03 11:43

<sup>1)</sup> A single subject may have reported medical history/concurrent diseases by more than one primary SOC category.

Table 5-3: Subjects reporting medical history/concurrent diseases and number of conditions by MedDRA System Organ Class (SOC) in Group B, Safety population

| | | | Restyla<br>N | | | | | Control<br>N = xx | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Primary SOC | | T | otal | Ongoing at study start | | | | Т | otal | 0 | ngoing a | t study start |
| | Su | bjects | Conditions | Subjects Conditions | | Subje | ects | Conditions | Subje | ects | Conditions | |
| | n | % | n | n | % | n | n | % | n | n | % | n |
| Total (N) <sup>1)</sup> | | | | | | | | | | | | |

<sup>% =</sup> n/N\*100

Version: 1.0 Effective date: 2017-11-03 11:43

<sup>1)</sup> A single subject may have reported medical history/concurrent diseases by more than one primary SOC category.

Effective date: 2017-11-03 11:43

SAP, 43CH1626, Restylane Volyme Midface

Doc id

Print date:

**MA-35135** 

Table 5-4: Prior use of facial fillers or implants, Safety population

| | | ( | Smorting V | | | Gro | ир В | | |
|---|---|---|---|---|---|---|---|---|---|
| Fillers/implants | Group A<br>N = xx | | | | • | rlane Volyme<br>N = xxx | Control<br>N = xx | | |
| | Sub | jects | Filers/implants | Sub | jects | Fillers/implants | Sub | jects | Fillers/implants |
| | n | % | n | n % | | n | n | % | n |
| Hyaluronic Acid (HA) | | | | | | | | | |
| Permanent implant | | | | | | | | | |
| Semi-permanent implant | | | | | | | | | |
| Collagen | | | | | | | | | |
| Other <sup>1)</sup> | | | | | | | | | |
| Total <sup>2)</sup> | | | | | | | | | |

<sup>% =</sup> n/N\*100

Table 5-5: Prior use of other facial dermatological procedures, Safety population

| | | <u></u> | Λ | | | Gro | ир В | | |
|---|---|---|---|---|---|---|---|---|---|
| Procedure | | | oup A | F | - | ne Volyme<br>= xxx | Control<br>N = xx | | |
| | Subjects Procedures | | Sub | jects | Procedures | Sub | jects | Procedures | |
| | n | % | n | n | % | n | n | % | n |
| Botulinum toxin injection | | | | | | | | | |
| Resurfacing | | | | | | | | | |
| Mesotherapy | | | | | | | | | |
| Face-lift | | | | | | | | | |
| Autologous Fat transplantation | | | | | | | | | |
| Other <sup>1)</sup> | | | | | | | | | |
| Total <sup>2)</sup> | | | | | | | | | |

<sup>% =</sup> n/N\*100

<sup>1)</sup> Specification of Other: ..., ....

<sup>2)</sup> A single subject may have had several fillers of implants.

<sup>1)</sup> Specification of Other: ..., ...,

<sup>2)</sup> A single subject may have had several facial dermatological procedures.

Print date:

2022-12-09 10:56

# 6 Appendix A3: Concomitant medication and procedures

### 6.1 Concomitant medication

Table 6-1: Subjects reporting concomitant medication, Safety population

| | Any concomitant medication | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Cra | A | | Group B | | | | | | | |
| Concomitant medication | | | up A<br>= xx | | Restylane Volyme N = xxx | | | | | | Control<br>N = xx | |
| | N | 0 | Y | es | No Yes | | No | | Yes | | | |
| | n | % | n | % | n | % | n | % | n | % | n | % |
| Ongoing at study start | | | | | | | | | | | | |
| Initiated during study | | | | | | | | | | | | |
| Total <sup>1)</sup> | | | | | | | | | | | | |

<sup>% =</sup> n/N\*100

Table 6-2: Subjects reporting concomitant medication and number of medications by reason, Safety population

| | | | Group A | ^ | | | | Gro | up B | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N = xx | | | | | Rest | ylane Vo<br>N = xxx | - | | Control<br>N = xx | | |
| Reason for concomitant medication | Sub | jects | | mber of dications | Sub | jects | Nu | mber of dications | Sub | jects | Nι | umber of dications |
| | n % Total at stu | | Ongoing<br>at study<br>end | n | % | Total | Ongoing<br>at study<br>end | n | % | Total | Ongoing<br>at study<br>end | |
| Related Adverse<br>Event | | | | | | | | | | | | |
| Unrelated<br>Adverse Event | | | | | | | | | | | | |
| Medical History | | | | | | | | | | | | |
| Other | | | | | | | | | | | | |
| Total <sup>1)</sup> | | | | | | | | | | | | |

<sup>% =</sup> n/N\*100

<sup>1)</sup> A single subject might have had concomitant medication ongoing at study start and initiated during study.

<sup>1)</sup> A single subject may have reported concomitant medication for several reasons.

2022-12-09 10:56

Print date:

Table 6-3: Subjects reporting concomitant medication and number of medications by ATC code, Safety population

| | | | <u></u> | oup A | | | Gro | ир В | | |
|---|---|---|---|---|---|---|---|---|---|---|
| ATC code | ATC text | | | oup A<br>= xx | F | | ine Volyme<br>= xxx | | | ontrol<br> = xx |
| Code | | Sub | jects | Medications | Sub | jects | Medications | Sub | jects | Medications |
| | | n | % | n | n | % | n | n | % | n |
| Total <sup>1)</sup> | | | | | | | | | | |

<sup>% =</sup> n/N\*100

Table 6-4: Subjects reporting concomitant medication taken due to an AE by ATC cod in Group A, Safety population

| | Concomitant medication | | | | |
|---|---|---|---|---|---|
| ATC and | ATO 1 1 | Subjects | Medications | PT | Related<br>AE |
| ATC code | ATC text | n | n | FI | |
| | | | | | Yes/No |
| | | | | | Yes/No |
| | | | | | Yes/No |
| | | | | | Yes/No |
| Total <sup>1)</sup> | | | | | |

<sup>% =</sup> n/N\*100

Note: if too much data for unrelated AEs then update this and the next table for related AEs only.

Table 6-5: Subjects reporting concomitant medication taken due to an AE by ATC code in Group B, Safety population

| | Concomitant medication | | | Adverse | e Event |
|---|---|---|---|---|---|
| ATO I- | ATC text | Subjects | Medications | PT | Related<br>AE |
| ATC code | ATC text | n | n | FI | |
| | | | | | Yes/No |
| | | | | | Yes/No |
| | | | | | Yes/No |
| | | | | | Yes/No |
| Total <sup>1)</sup> | | | | | |

<sup>% =</sup> n/N\*100

<sup>1)</sup> A single subject may have reported several types of concomitant medication.

<sup>1)</sup> A single subject may have reported several types of concomitant medication.

<sup>1)</sup> A single subject may have reported several types of concomitant medication.

Doc id SAP, 43CH1626, Restylane Volyme Midface ♣ GALDERMA **MA-35135** 

Print date:

2022-12-09 10:56

#### **6.2 Concomitant procedures**

Table 6-6: Subjects reporting concomitant procedures and number of procedures by reason, Safety population

| | | Group A | | | Group B | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Reason for concomitant | N = xx | | | Restylane Volyme<br>N = xxx | | | Control<br>N = xx | | |
| procedure | Sub | jects | ts Procedures | | Subjects Procedures | | Subjects | | Procedures |
| | n | % | n | n | % | n | n | % | n |
| Adverse Event | | | | | | | | | |
| Medical History | | | | | | | | | |
| Other | | | | | | | | | |
| Total <sup>1)</sup> | | | | | | | | | |

<sup>% =</sup> n/N\*100

Please consider to add a table regarding "Concomitant procedures due to a related AE".

Table 6-7: Subjects reporting concomitant procedures and number of procedures, Safety population

| | Group A | | Group B | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Concomitant procedure | N = xx | | | Restylane Volyme<br>N = xxx | | | Control<br>N = xx | | |
| | Subjects Procedures | | Subjects Procedures | | Subjects Procedure | | Procedures | | |
| | n | % | n | n | % | n | n | % | n |
| Total <sup>1)</sup> | | | | | | | | | |

<sup>% =</sup> n/N\*100

Note: if too much data for unrelated AEs then update this table for related AEs only.

<sup>1)</sup> A single subject may have reported procedures for several reasons.

<sup>1)</sup> A single subject may have reported several concomitant procedures.

SAP, 43CH1626, Restylane Volyme Midface Doc id ♣ GALDERMA MA-35135

#### Appendix A4: Treatment procedure 7

Table 7-1: Exposure to study treatment, Safety population

| | Parameter | One A | Group B | |
|---|---|---|---|---|
| Assessment (right and left midface combined) | | Group A<br>N = xx | Restylane Volyme<br>N = xxx | Control<br>N = xx |
| Volume injected (mL) at initial treatment | N | | | |
| | Mean (SD) | | | |
| | Median | | | |
| | Minimum,<br>Maximum | | | |
| Volume injected (mL) at touch-up | N | | | |
| | Mean (SD) | | | |
| | Median | | | |
| | Minimum,<br>Maximum | | | |
| Total volume injected (mL) at initial treatment and touch-up | N | | | |
| | Mean (SD) | | | |
| | Median | | | |
| | Minimum,<br>Maximum | | | |
| Depth of injection at initial treatment | | | | |
| Subcutaneous | n (%) | | | |
| Supraperiosteal | n (%) | | | |
| Other <sup>1)</sup> | n (%) | | | |
| Depth of injection at touch-up | | | | |
| Subcutaneous | n (%) | | | |
| Supraperiosteal | n (%) | | | |
| Other <sup>2)</sup> | n (%) | | | |
| Injection method at initial treatment | | | | |
| Linear retrograde | n (%) | | | |
| Small aliquots | n (%) | | | |
| Fanning injection technique | n (%) | | | |
| Other <sup>3)</sup> | n (%) | | | |

Doc id

Print date:

MA-35135

2022-12-09 10:56

| A | | Croup A | Group B | |
|---|---|---|---|---|
| Assessment (right and left midface combined) | Parameter | Group A<br>N = xx | Restylane Volyme<br>N = xxx | Control<br>N = xx |
| Injection method at touch-up | | | | |
| Linear retrograde | n (%) | | | |
| Small aliquots | n (%) | | | |
| Fanning injection technique | n (%) | | | |
| Other4) | n (%) | | | |

<sup>% =</sup> n/N\*100

Effective date: 2017-11-03 11:43

<sup>1)</sup> Specification of Other: ..., ...,

<sup>2)</sup> Specification of Other: ..., ...,

<sup>3)</sup> Specification of Other: ..., ...,

<sup>4)</sup> Specification of Other: ..., ..., ....

Effective date: 2017-11-03 11:43

SAP, 43CH1626, Restylane Volyme Midface

Doc id

Print date:

MA-35135

2022-12-09 10:56

Table 7-2: Treatment procedure, Safety population

| Accessment /::-l-t | | | | Group B | |
|---|---|---|---|---|---|
| Time<br>Point | Assessment (right and left midface combined) | Category | Group A<br>N = xx | Restylane Volyme<br>N = xxx | Control<br>N = xx |
| | , | | | n (%) | n (%) |
| Initial<br>treatment | Local anaesthesia used? | No | | | |
| | | Yes | | | |
| | | Whereof topical cream | | | |
| | | Whereof local infiltration | | | |
| Touch-up | Local anaesthesia used? | No | | | |
| | | Yes | | | |
| | | Whereof topical cream | | | |
| | | Whereof local infiltration | | | |
| Initial<br>treatment | Post-treatment care | None | | | |
| | | Massage | | | |
| | | Ice pack | | | |
| | | Other <sup>1)</sup> | | | |
| Touch-up | Post-treatment care | None | | | |
| | | Massage | | | |
| | | Ice pack | | | |
| | | Other <sup>1)</sup> | | | |

<sup>% =</sup> n/N\*100

Any device deficiencies will be listed in text or in a separate table, as appropriate.

<sup>1)</sup> Specification of Other: ..., ...,

<sup>2)</sup> Specification of Other: ..., ...,

# 8 Appendix A5: Post-treatment examinations

Table 8-1: Subjects with change from baseline in post-treatment BMI ≥ 2 units, Safety population

| Group | A | Group B | |
|---|---|---|---|
| Number of subjects | Subject numbers | Number of subjects | Subject numbers |
# Appendix A6: Effectiveness Evaluation for Group B 9

# 9.1 Primary analysis

## 9.1.1 MMVS responder rate at Month 6

Table 9-1: MMVS responder rate at Month 6 by treatment, Blinded Evaluator

| Population | Assessment/Time Point | Treatment group | Subjects in population | Respo | nders | 95% Confidence Interval | P-value |
|---|---|---|---|---|---|---|---|
| | | | N | n | % | | |
| FAS <sup>1)</sup> | Right and left midface combined at Month 6 | Restylane Volyme | | | | | |
| | | Control | | | | | |
| | | Difference | | | | | |
| PP <sup>2)</sup> | Right and left midface combined at Month 6 | Restylane Volyme | | | | | |
| | | Control | | | | | |
| | | Difference | | | | | |

<sup>1)</sup> Subjects with a missing MMVS score have their values imputed using BOCF up to Month 6.

Note: Responder rate (%) = n/N\*100

Page 36 of 63

<sup>2)</sup> No imputation is used for PP analysis. Only subjects with complete data are included.

Note: Responder is defined as a subject with an improvement of at least one grade on the MMVS from baseline.

GALDERMA SAP, 43CH1626, Restylane Volyme Midface

MA-35135

Doc id



SAP, 43CH1626, Restylane Volyme Midface

Doc id

Print date:

MA-35135

2022-12-09 10:56

Effective

SAP, 43CH1626, Restylane Volyme Midface

MA-35135

Doc id



Print date: 2022-12-09 10:56

GALDERMA

Title
SAP, 43CH1626, Restylane Volyme Midface

MA-35135







SAP, 43CH1626, Restylane Volyme Midface

MA-35135

2022-12-09 10:56

Print date:

Doc id

CCI



Effective date: 2017-11-03 11:43

Effective

SAP, 43CH1626, Restylane Volyme Midface

MA-35135

2022-12-09 10:56

Print date:

Doc id

Effective

Version: 1.0

SAP, 43CH1626, Restylane Volyme Midface

MA-35135

2022-12-09 10:56

Print date:

Doc id

Print date: 2022-12-09 10:56

GALDERMA

Table
SAP, 43CH1626, Restylane Volyme Midface

MA-35135

• GALDERMA SAP,

SAP, 43CH1626, Restylane Volyme Midface

Doc id

Print date:

MA-35135

2022-12-09 10:56

Effective

GALDERMA

Title SAP, 43CH1626, Restylane Volyme Midface

MA-35135





SAP, 43CH1626, Restylane Volyme Midface

2022-12-09 10:56

Print date:

Doc id

MA-35135

SAP, 43CH1626, Restylane Volyme Midface Doc id 👶 GALDERMA MA-35135

| CCI |
|-----|

GALDERMA

Title SAP, 43CH1626, Restylane Volyme Midface

MA-35135

| CCI |
|-----|





Effective

Version: 1.0

SAP, 43CH1626, Restylane Volyme Midface

Doc id

Print date:

MA-35135

2022-12-09 10:56

Effective

Version: 1.0

SAP, 43CH1626, Restylane Volyme Midface

Doc id

Print date:

MA-35135

2022-12-09 10:56

SAP, 43CH1626, Restylane Volyme Midface

MA-35135

2022-12-09 10:56

Print date:

Doc id

Effective

Doc id SAP, 43CH1626, Restylane Volyme Midface ♣ GALDERMA MA-35135

# **Appendix A7: Safety evaluation 10**



GALDERMA

Title
SAP, 43CH1626, Restylane Volyme Midface

MA-35135



GALDERMA

Title SAP, 43CH1626, Restylane Volyme Midface

MA-35135

| CCI |
|-----|

SAP, 43CH1626, Restylane Volyme Midface

Doc id

Print date:

**MA-35135** 

2022-12-09 10:56

# **Adverse Events** 10.2

### 10.2.1 Summary of Adverse Events (AEs)

Table 10-5: Brief summary of all AEs, Safety population

| | | | | | | Grou | ир В | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Group<br>N = x | | No | treatm<br>baseli<br>N = x | | Treatmer<br>Restylane<br>N = x | | Volyme |
| | Sub | jects | Events | Subjects | | Events | Subjects | | Events |
| | n | % | n | n | % | n | n | % | n |
| Any AEs reported, total | | | | | | | | | |
| AEs related to product and/or injection procedure | | | | | | | | | |
| Of which were serious | | | | | | | | | |
| AEs unrelated to product and/or injection procedure | | | | | | | | | |
| of which were serious | | | | | | | | | |
| Subjects with no AE reported | | | | | | | | | |

<sup>% =</sup> n/N\*100

Note: Treatment with Restylane Volyme columns include data from subjects in the Restylane Volyme group after their initial treatment at baseline, as well as data from subjects in the Control group after their initial treatment at Month 6.

Doc id SAP, 43CH1626, Restylane Volyme Midface ♣ GALDERMA MA-35135

Print date:

2022-12-09 10:56

#### 10.2.2 Related AEs

Table 10-6: Related AEs occurring throughout the whole study period by MedDRA System Organ Class, Preferred Term, and maximum intensity, Safety population, Group B

| Primary System<br>Organ Class | Maximum | No treatn<br>basel<br>N = | ine | Treatme<br>Restylane<br>N = 2 | Volyme | To<br>N = | |
|---|---|---|---|---|---|---|---|
| Preferred Term | intensity | Subjects | Events | Subjects | Events | Subjects | Events |
| | | n (%) | n | n (%) | n | n (%) | n |
| Any related AE | Total | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| SOC1 | Total | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| PT11 | Total | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| PT12 | Total | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| SOC2 | Total | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| PT21 | Total | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| % = n/N*100 | 1 | I | 1 | | l | 1 | |

<sup>% =</sup> n/N\*100

Note: Treatment with Restylane Volyme columns include data from subjects in the Restylane Volyme group after their initial treatment at baseline, as well as data from subjects in the Control group after their initial treatment at Month 6.

Table 10-7: Duration (number of days days) of related AEs occurred throughout the whole study period by MedDRA System Organ Class and Preferred Term, Safety population, Group B

| Primary<br>System Organ<br>Class | No treatment at baseline<br>N = xx | | | Treatment with Restylane Volyme N = xxx | | | | Total<br>N = xxx | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred<br>Term | N<br>(events) | Duration missing | Mean<br>(SD) | Median | Min-<br>Max | N<br>(events) | Duration missing | Mean<br>(SD) | Median | Min-<br>Max | N<br>(events) | Duration missing | Mean<br>(SD) | Median | Min-<br>Max |
| SOC1 | | | | | | | | | | | | | | | |
| PT11 | | | | | | | | | | | | | | | |
| PT12 | | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | | |

Note: Treatment with Restylane Volyme columns include data from subjects in the Restylane Volyme group after their initial treatment at baseline, as well as data from subjects in the Control group after their initial treatment at Month 6.

Table 10-8: Time to onset (days) since most recent treatment of related AEs by MedDRA System Organ Class and Preferred Term, Safety population, Group B

| | No treatment at baseline | | | | Treatment with Restylane Volyme | | | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Primary System Organ<br>Class | N = xx | | | | N = xxx | | | | N = xxx | | | |
| Preferred Term | N<br>(events) | Mean (SD) | Median | Min-Max | N<br>(events) | Mean (SD) | Median | Min-Max | N<br>(events) | Mean (SD) | Median | Min-Max |
| SOC1 | | | | | | | | | | | | |
| PT11 | | | | | | | | | | | | |
| PT12 | | | | | | | | | | | | |
| Total | | | | | | | | | | | | |

Note: Treatment with Restylane Volyme columns include data from subjects in the Restylane Volyme group after their initial treatment at baseline, as well as data from subjects in the Control group after their initial treatment at Month 6.

**Effective** 

Version: 1.0

GALDERMA

Title
SAP, 43CH1626, Restylane Volyme Midface

MA-35135

Table 10-9: Action taken due to related AEs by MedDRA System Organ Class and Preferred Term, Safety population

| | | | | | | Ac | tion Taken | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System | | No tre | eatment at baseline | | Treatment with Restylane Volyme | | | | | Total | | |
| Organ | | | N = xx | | N = xxx | | | | | | N = xxx | |
| Class<br>Preferred<br>Term | None | Medication treatment | Non-<br>pharmacological<br>treatment or<br>other<br>procedures/tests | Subject<br>withdrawn | None | Medication treatment | Non-<br>pharmacological<br>treatment or<br>other<br>procedures/tests | Subject<br>withdrawn | None | Medication treatment | Non-<br>pharmacological<br>treatment or<br>other<br>procedures/tests | Subject<br>withdrawn |
| SOC 1 | | | | | | | | | | | | |
| PT11 | | | | | | | | | | | | |
| PT12 | | | | | | | | | | | | |
| SOC 2 | | | | | | | | | | | | |
| PT21 | | | | | | | | | | | | |
| PT22 | | | | | | | | | | | | |
| All | | | | | | | | | | | | |

Note: Treatment with Restylane Volyme columns include data from subjects in the Restylane Volyme group after their initial treatment at baseline, as well as data from subjects in the Control group after their initial treatment at Month 6.

Effective

Doc id SAP, 43CH1626, Restylane Volyme Midface ♣ GALDERMA **MA-35135** 

Print date:

2022-12-09 10:56

#### 10.2.3 Unrelated AEs

Table 10-10: Unrelated AEs by MedDRA System Organ Class, Preferred Term, and maximum intensity, Safety population

| Primary System<br>Organ Class | Maximum | No treatr<br>basel<br>N = | line | Treatme<br>Restylane<br>N = | Volyme | To<br>N = | |
|---|---|---|---|---|---|---|---|
| Preferred Term | intensity | Subjects | Events | Subjects | Events | Subjects | Events |
| | | n (%) | n | n (%) | n | n (%) | n |
| Any related AE | Total | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| SOC1 | Total | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| PT11 | Total | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| PT12 | Total | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| SOC2 | Total | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| PT21 | Total | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| $\frac{0}{0} = n/N*100$ | I | l | 1 | | L | 1 | |

<sup>% =</sup> n/N\*100

Note: Treatment with Restylane Volyme columns include data from subjects in the Restylane Volyme group after their initial treatment at baseline, as well as data from subjects in the Control group after their initial treatment at Month 6.

ERMA
Title
SAP, 43CH1626, Restylane Volyme Midface
MA-35135

Print date:

2022-12-09 10:56

# SIGNATURES PAGE

| Date | Signed by |
|------------------|------------------------------|
| 2017-11-01 17:09 | PPD |
| Justification | Approved by Technical Expert |
| 2017-11-02 08:19 | PPD |
| Justification | Approved by Technical Expert |
| 2017-11-02 14:06 | PPD |
| Justification | Approved by Technical Expert |
| 2017-11-03 05:42 | PPD |
| Justification | Approved by Technical Expert |
| | ' |
| 2017-11-03 11:43 | PPD |
| Justification | Approved by Owner |